CLINICAL TRIAL: NCT04583722
Title: Clinical Evaluation of a New Encapsulation Technology for Improving Astaxanthin Bioavailability Based on Natural Food Ingredients Only
Brief Title: Evaluating Astaxanthin Bioavailability, and a New Technology for Improving it, Using Natural Food Materials Only
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yoav D. Livney (Other)
Collaborators: Israel Innovation Authority (Unknown)
Responsible Party: Sponsor-Investigator, Yoav D. Livney, Prof., Technion, Israel Institute of Technology
Organization: Technion, Israel Institute of Technology (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 0048-18-RMB
Record Dates: First submitted 2020-10-05; First posted 2020-10-12 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Bioavailability
Keywords: Astaxanthin; Bioavailability; Encapsulation; Potato protein; Olive oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AX oleoresin (Other): Raw AX oleoresin, 15 mg AX (in 4 pululan capsules)
  Interventions: Dietary Supplement: AX-olive oil-PP emulsion
- AX-olive oil-PP emulsion (Experimental): Microencapsulated AX (1%:2%:3% (AXO:OO:PP, %w/v ratio) + 0.15% maltodextrin). 15 mg AX (in 4 pululan capsules)
  Interventions: Dietary Supplement: AX-olive oil-PP emulsion

INTERVENTIONS:
Dietary Supplement: AX-olive oil-PP emulsion — single dose and plasma samples
  Other Names: (control- raw AXoleoresin)

SUMMARY:
The purpose of this study was to develop a potato protein (PP)-based delivery system for increasing oral bioavailability of lipophilic bioactives (nutraceuticals and drugs), using astxanthin (AX) as a model, and to evaluate the system in vivo in a crossover clinical study in human volunteers. Three different formulations were prepared, encapsulating AX oleoresin (AXO) with (1) PP only, (2) PP+lecithin (LEC), and (3) PP+olive oil (OO). In a randomized, double-blind, crossover study in human subjects, the PP-OO-AX formulation had a 4.8-fold higher median plasma AX area under the concentration-over time curve (AUC; P<0.001) compared to the raw AXO formulation.

In conclusion, a non-allergenic, vegan, PP based delivery system made of "all-natural ingredients" offers a great promise for increasing oral bioavailability of lipophilic bioactives such as AX, for the enrichment of food and for dietary supplements, or oral delivery of lipophilic drugs.

DETAILED DESCRIPTION:
Astaxanthin (AX) is a red xanthophyll carotenoid found mainly in algae (notably Haematococcus Pluvialis microalga) and marine animals. AX is a stronger antioxidant than vitamin E and β-carotene but has very low oral bioavailability. The purpose of this study was to develop a potato protein (PP)-based delivery system for increasing oral bioavailability of lipophilic bioactives (nutraceuticals and drugs), using AX as a model, and to evaluate the system in vitro and in vivo in a crossover clinical study in human volunteers. Three different formulations were prepared, encapsulating AX oleoresin (AXO) with (1) PP only, (2) PP+lecithin (LEC), and (3) PP+olive oil (OO). The average particle diameters after preparation were 0.29, 0.29, and 1.76 μm, and after freeze-drying and reconstitution 0.17, 0.07, and 6.93 μm, respectively. In vitro bioaccessibility was 33, 47, and 69%, respectively, versus 16% only for the raw AXO. In a randomized, double-blind, crossover study in human subjects, the PP-OO-AX formulation had a 4.8-fold higher median plasma AX area under the concentration-over time curve (AUC; P<0.001) compared to the raw AXO formulation. In conclusion, a non-allergenic, vegan, PP based delivery system made of "all-natural ingredients" offers a great promise for increasing oral bioavailability of lipophilic bioactives such as AX, for the enrichment of food and for dietary supplements, or oral delivery of lipophilic drugs.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Aged 18 - 26
* Normal physical examination
* Normal electrocardiogram (E.C.G.)
* Normal laboratory profile

Exclusion Criteria:

* Any active medical illness (e.g. liver disease, kidney disease, or diabetes, intestinal malabsorption, hypercalcemia)
* Lactose intolerance
* Food allergies
* Excessive alcohol use (over 40 ml/day)
* Pregnant or breast-feeding
* Hyperlipidemia (LDL>130, triglycerides>200)
* Regular medication use
* Obesity (BMI>30 kg/m2)
* Use of multivitamins, or carotenoid supplements during the past month prior to the study
* Current smoking

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2018-07-15 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-01-16 (Actual)

PRIMARY OUTCOMES:
Plasma AX AUC | 1 year
  Plasma AX AUC of 13 participants after consuming either the microencapsulated AX or the reference AX oleoresin, measured during 72 hrs post-ingestion, in a cross over study.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Segal, Doctor, Principal Investigator — Endocrine Institute, Rambam Health Care Campus
Locations (1):
- Rambam Health Campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abuhassira-Cohen Y, Edelman R, Abbas R, Kurnik D, Shibel R, Livney YD, Enhancing the oral bioavailability of natural astaxanthin using plant-based micro- and nano-encapsulation materials: Results of an In vitro evaluation and a cross-over study in humans, Precision Nanomedicine 2020; 3 (4), 641-655.
- See also: The publication reporting the clinical study — https://doi.org/10.33218/001c.16781